CLINICAL TRIAL: NCT07355907
Title: Comparison of Preoperative Prophylactic Single Dose Fosfomycin Trometamol Versus 5-day Levofloxacin in Prevention of Post-percutaneous Nephrolithotomy Infectious Complications and Sepsis: A Prospective Randomized Controlled Trial.
Brief Title: Preoperative Prophylactic Fosfomycin Trometamol Versus 5-day Levofloxacin in Prevention of Postpercutaneous Nephrolithotomy Infectious Complications and Sepsis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Zoeir, Tanta, ElGeish street, Gharbiya government, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35524/6/22
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Calculi, Renal; PCNL; Infectious Complications
Keywords: renal stones; PCNL; INFECTION; SEPSIS; ANTIBIOTIC PROPHYLAXIS
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Infections; Sepsis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preoperative Fosfomycin Trometamol group (Active Comparator): Fosfomycin before PCNL
  Interventions: Procedure: PCNL
- Preoperative 5-day Levofloxacin group (Active Comparator): Levofloxacin before PCNL
  Interventions: Procedure: PCNL
- No preopertive antibiotic group (Other): control, no preoperative antibiotic before PCNL
  Interventions: Procedure: PCNL

INTERVENTIONS:
Procedure: PCNL — PCNL for renal stones

SUMMARY:
A randomized controlled trial comparing the use of preoperative prophylactic single dose fosfomycin trometamol versus levofloxacin in prevention of post-PCNL infectious complications and sepsis.

the 3 groups were compared as regards the baseline data, preoperative data, intra-operative data, and post-op data.

DETAILED DESCRIPTION:
A prospective randomized study, in which 300 patients admitted to urology department, Tanta university with renal stones prepared for PCNL were randomly distributed into 3 groups:

Group I, included 70 patients received single oral dose Fosfomycin 3 gm the night before the procedure.

Group II, included 70 patients received 5 days levofloxacin 500 mg once daily before PCNL Group III, included 70 patients will not receive preoperative treatment

The patients were evaluated by: complete hemogram, renal function, stone work-up, and MSU culture were done preoperatively.

NCCT was done for all included patients Intraoperative renal pelvic urine (collected after ureteral catheterization or at first puncture of pelvicalyceal system [PCS]) and stone fragments were collected in sterile plastic containers for culture. The samples were sent immediately (within 1 hour) to the laboratory for processing.

The following data were recorded and compared; patients' demographic data, stone characteristics, preoperative lab. Investigations, intraoperative data (OR time and complications) and postoperative data (SFR, complications especially infectious ones, sepsis and fever, hospital stay), and post-operative bacteruria.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with renal stones scheduled for PCNL

Exclusion Criteria:

* Unfit patients for surgery
* patients with active UT
* uncorrected coagulopathy
* pregnancy
* children

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
post-operative infectious complications and sepsis | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided